CLINICAL TRIAL: NCT06886490
Title: Effects of Plant-based Diets on Body Weight and Selected Metabolic Parameters in Obese Patients: a Randomised Controlled Trial of Five Different Diets
Brief Title: Plant-based Diets and Body Weight and Selected Metabolic Parameters Management in Obese Patients.
Acronym: VEGPREV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, ANNA JAGIELSKA, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB/37/2023
Record Dates: First submitted 2025-02-18; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-01

CONDITIONS: Obesity and Overweight; Dietary Intervention; Vegetarian Diet; Vegan Diet; Mediterranean Diet; Metabolic Cardiovascular Syndrome
Keywords: Dietary intervention; plant-based diets; Obesity and overweight; randomised controlled trial
MeSH Terms: conditions — Obesity; Overweight; Metabolic Syndrome | interventions — Diet, Mediterranean; Diet, Vegetarian; Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Mediterranean diet (Experimental): This heart-healthy eating plan emphasizes healthy fats, whole grains, fruits, vegetables, beans, nuts and seeds.
  Interventions: Other: Mediterranean diet
- Planetary diet (Experimental): Defined in the EAT-Lancet Commission report
  Interventions: Other: Planetary diet
- Lactovegetarian diet (Experimental): A variation of vegetarianism that excludes meat, poultry, seafood, and eggs, but includes dairy products.
  Interventions: Other: Lactovegetarian diet
- Vegan diet (Experimental): Based on plants (such as vegetables, grains, nuts and fruits) and foods made from plants.
  Interventions: Other: Vegan diet
- Control diet (Experimental): Based on the current national dietary recommendations for the Polish population
  Interventions: Other: Control diet

INTERVENTIONS:
Other: Mediterranean diet — VEGPREV study is a randomized intervention trial with an intervention period of 12 weeks, and follow-up after another 12-14 weeks conducted at the Department of Social Medicine and Public Health at Warsaw Medical University. Study aim is to evaluate the efficacy of the following plant-based diet: Mediterranean diet: Animal : vegetable protein ratio - 70:30.
  Arms: Mediterranean diet
Other: Planetary diet — VEGPREV study is a randomized intervention trial with an intervention period of 12 weeks, and follow-up after another 12-14 weeks conducted at the Department of Social Medicine and Public Health at Warsaw Medical University. Study aim is to evaluate the efficacy of the following plant-based diet: Planetary diet: Reduce consumption of red meat, moderate consumption of poultry, fish and seafood and their products, and eggs and dairy. Animal : vegetable protein ratio - 50:50
  Arms: Planetary diet
Other: Lactovegetarian diet — VEGPREV study is a randomized intervention trial with an intervention period of 12 weeks, and follow-up after another 12-14 weeks conducted at the Department of Social Medicine and Public Health at Warsaw Medical University. Study aim is to evaluate the efficacy of the following plant-based diet: Lactovegetarian diet: Reduce consumption of meat, fish and seafood and their preparations, and eggs and dairy products. Animal : vegetable protein ratio - 30:70.
  Arms: Lactovegetarian diet
Other: Vegan diet — VEGPREV study is a randomized intervention trial with an intervention period of 12 weeks, and follow-up after another 12-14 weeks conducted at the Department of Social Medicine and Public Health at Warsaw Medical University. Study aim is to evaluate the efficacy of the following plant-based diet: Vegan diet: Excludes all animal and animal-derived products (meat, fish, seafood, dairy, eggs, honey).
  Arms: Vegan diet
Other: Control diet — VEGPREV study is a randomized intervention trial with an intervention period of 12 weeks, and follow-up after another 12-14 weeks conducted at the Department of Social Medicine and Public Health at Warsaw Medical University. Study aim is to evaluate the efficacy of the following plant-based diet: Control diet: Reduce consumption of red meat, consumption of poultry, fish and seafood and their products, regular consumption of eggs and dairy products.
  Arms: Control diet

SUMMARY:
The aim of the study is to determine the optimal plant-based dietary model in terms of weight loss and health that would be both acceptable and environmentally friendly dietary model based on limiting the consumption of meat and animal products. Such findings will lead to new knowledge and allow us to formulate new principles for the nutritional treatment of people suffering from obesity.

DETAILED DESCRIPTION:
Obesity is not only one of the most serious health problems in the world, it is also associated with an increased risk of many other diseases. Despite many preventive measures, the number of people suffering from obesity is constantly increasing, also in Poland. One of the integral elements of treatment is a change in lifestyle, including a change in eating habits. In this context, new dietary models are constantly being considered and eagerly adopted by patients. These are not always rational and evidence-based choices. What's more, what we eat is not only important for our health, but also for the planet. Recently, high-fat diets with a significant carbon footprint have gained popularity.

It is therefore worth considering more plant-based dietary models in the treatment of obesity and its associated disorders. Such a change can simultaneously help reduce greenhouse gas emissions and improve environmental quality, as well as benefit our health - both directly and indirectly.

There is a growing body of scientific evidence suggesting that limiting meat consumption may be beneficial to health, leading to weight loss, improvements in selected cardiovascular risk parameters and inflammation. However, many questions remain.

For this reason, more plant-based dietary patterns are worth considering in the treatment of obesity and its accompanying disorders. There is growing scientific evidence that limiting meat consumption promotes good health. It has been shown that the implementation of a vegetarian diet can result in weight loss, as well as help in maintaining optimal weight levels more effectively in the long term. This is extremely important for people suffering from obesity. Adherence to meat-restricted diets is also associated with other health benefits, which include an improved lipid profile and other cardiovascular risk parameters, as well as beneficial effects on inflammation and oxidative stress parameters.

Currently, there are only a few intervention studies available that have investigated the effectiveness of plant-based diets in a population of obese adults who previously have not restricted their meat consumption. Most of the studies concern vegetarians, whose awareness of taking care of their diet and lifestyle is, after all, much higher. To some extent, this may explain such optimistic conclusions from observational studies. It is not the only issue associated with research focused on plant-based diets. In experimental studies, the results of dietary interventions are very often compared with no intervention whatsoever. It would therefore be interesting to verify the effectiveness of a vegan or vegetarian diet against current dietary recommendations or another health-promoting dietary pattern - the Mediterranean diet. After all, vegan or vegetarian diets are elimination diets. Should they be recommended for the treatment of obesity and disorders associated with it? Do body weight, cholesterol and glucose levels decrease faster? What risks do they entail and are they difficult to implement? The investigators only know the answers to some of these questions.

In light of the above facts, the study will aim to evaluate the efficacy of the following plant-based diets: (1) the Mediterranean diet, (2) the 'planetary diet' as defined in the EAT-Lancet Commission report (3), the lactovegetarian diet, and (4) the vegan diet, in terms of weight reduction and effects on selected metabolic factors among obese patients. The last group (5) will receive the current national dietary recommendations for the Polish population.

To the investigators best knowledge, this is the first such study in Poland comparing several different plant-based diets. The investigators plan to recruit 100 obese adults under 60 years of age. The cohort will be randomly divided into five groups, each receiving a different intervention for 12 weeks. After 12 to 14 weeks from the end of the intervention, a follow-up meeting will take place again (i.e. after 24 to 26 weeks from the start of the nutritional intervention).

The study collect socio-demographic data and information on lifestyle (including dietary habits, physical activity, substance use and diet supplementation), psychological questionnaires (Perception of their own ability to change their diet (personality resources), which will be determined by the intensity of self-efficacy (GSES scale); Positive attitude towards the future, which will be determined by assessing the intensity of optimism (LOT-R); Coping dealing with emotions, which will be determined by assessing emotional control (CECS emotional control scale); Human ability to respond flexibly to changing situation requirements (stress, conflict, uncertainty), which will be determined by use The Brief Resilience Coping Scale (BRCS) created by V. G. and K. Sinclair A. Wallston) and to carry out biochemical tests and anthropometric measurements. Patients will be given dietary recommendations appropriate to the diet and specially designed dietary schemes, the main element to be intervened upon being the frequency of consumption of meat and other animal products or their elimination. In addition, an average carbon footprint will be estimated for each diet. Meetings with the dietitian will take place in a hybrid format (face-to-face and on-line). Venous blood for biochemical testing will be collected from patients before and after the study and at week 6 of the intervention. At the same time, anthropometric measurements will also be taken and information on wellbeing or difficulties in meeting dietary recommendations will be recorded. The investigators plan to examine the effects of the intervention on changes in body weight, body composition, blood pressure and, among others, changes in total cholesterol, LDL fraction, HDL fraction, changes in triacylglycerols, blood glucose, insulin, reduction in blood uric acid or changes in ALT, AST, GGTP activity.

Also, biochemical tests will be performed, including tests for inflammatory parameters (C-reactive protein (CRP), interleukin-6 (IL-6), L-selectin, intercellular adhesion molecule-1 (ICAM-1), and adiponectin), as well as anthropometric measurements and body composition assessments based on electrical bioimpedance. TMAO concentrations will be examined in relation to selected appetite traits. In addition, metabolites and cofactors of the methionine cycle (S-(5'-Adenosyl)-L-homocysteine (SAH), homocysteine, methionine, S-(5'-Adenosyl)-L-methionine (SAM), choline, betaine) will be monitored. In addition, selected polymorphisms of genes related to the homocysteine-methionine cycle and lipid metabolism will be evaluated. Patients will be given dietary recommendations according to their dietary habits, with the frequency of consumption or elimination of meat and other zoonotic products and their products as the main intervention element. Meetings with the dietitian will be held at baseline, week 6 and week 12. Between meetings, weekly online visits with a psychodietitian will be scheduled.

The aim of the study is to determine the optimal dietary model in terms of weight loss and health that would be both acceptable and environmentally friendly dietary model based on limiting the consumption of meat and animal products. The goal of this study is also to evaluate the efficacy of selected plant-based diets on weight loss, effects on selected metabolic and inflammatory parameters in obese adults. Such findings will lead to new knowledge and allow us to formulate new principles for the nutritional treatment of people suffering from obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years (adults able to give informed consent to participate in the study) ≤ 60 years of age
* BMI >30 kg/m2 or BMI 25-29.9 kg/m2 with waist circumference in women 88 cm, in men 94cm.

Exclusion Criteria:

* age <18 years and >60 years,
* severe medical conditions, including alcoholism, major and extensive surgery, chronic kidney and liver disease, history of myocardial infarction, unstable angina pectoris within the last 6 months, history of stroke within the last 6 months, cancer within the last 5 years,
* psychiatric condition preventing participation in the study and cooperation with the investigators,
* use of enteral or parenteral nutrition,
* use of medications that cause significant weight loss (e.g., GLP-1 analogues)
* pregnancy or breast feeding,
* attempts to change dietary habits, including reduction of caloric intake and elimination of meat and animal products in the past 6 months,
* lack of consent to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Body weight | After 12 weeks of dietary intervention
  Mean incremental difference in body weight (kg) change of 1% consecutively between each of the five groups (corresponding to an effect size of 0.57)

SECONDARY OUTCOMES:
Waist and hip circumference | After 12 weeks of intervention
  Waist and hip circumference changes in cm.
Waist-Hip Ratio (WHR) | After 12 weeks of intervention
  Waist (in cm) and hip circumference (in cm) will be combined to report WHR changes.
Body fat mass | After 12 weeks of intervention]
  Body mass fat expressed in kg and as a percentage of body mass (%) changes.
Lipids profile | After 12 weeks of intervention
  Evaluation of lipid metabolism changes by: total cholesterol (mg/dl) , LDL - cholesterol (mg/dl), HDL - cholesterol (mg/dl), triacylglycerols (mg/dl) levels.
Glucose level changes | After 12 weeks of intervention.
  Assessment of metabolic changes related to glucose regulation by fasting glucose (in mg/dl).
Insulin level changes | After 12 weeks of intervention
  Assessment of metabolic changes related to glucose regulation by fasting insulin (in μIU/ml) levels.
Blood Uric Acid | After 12 weeks of intervention
  Evaluation of intervention effects on purine metabolism by blood uric acid (mg/dl) level change.
Serum Micronutrient Levels | After 12 weeks of intervention
  Changes in folic acid (ng/ml), ferritin (ng/ml), iron (μg/dl), and vitamin D3 (ng/ml) vitamin B12 (pg/ml) blood concentration to assess alterations in micronutrient levels in response to the intervention.
Liver Enzymes Activity | After 12 weeks of intervention
  Changes in ALT (U/l), AST (U/l), and GGTP (U/l) activity to assess liver function alterations.
Inflammatory Markers | After 12 weeks of intervention
  Changes in levels of CRP (mg/l), IL-6 (pg/mL), IL-18 (pg/mL), IL-1RA (pg/mL), E-selectin (ng/mL), ICAM-1 (ng/mL), MCP-1 (pg/mL), adiponectin (µg/mL), omentin-1 (ng/mL), and resistin (ng/mL) to analyse systemic inflammation responses.

OTHER OUTCOMES:
Methionine cycle metabolites and related compounds and Choline pathway metabolites. | After 12 weeks of intervention
  Changes in: S-(5'-Adenosyl)-L-homocysteine (SAH) (nmol/L), Homocysteine (µmol/L), Methionine (µmol/L), S-(5'-Adenosyl)-L-methionine (SAM) (nmol/L), Choline (µmol/L), Betaine (µmol/L) levels to evaluate changes in one-carbon metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Jagielska, MD, PhD, Principal Investigator — Medical University of Warsaw, Department od Social Medicine and Public Health
Locations (1):
- Department of Social Medicine and Public Health, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided